CLINICAL TRIAL: NCT05059769
Title: Relationship Between Ambulatory Arterial Stiffness Index and Left Ventricular Diastolic Function in Patients With HFpEF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dongying Zhang (Other)
Responsible Party: Sponsor-Investigator, Dongying Zhang, Clinical Professor, Chongqing Medical University
Organization: Chongqing Medical University (Other)
Other Study IDs: 2020-09-21
Record Dates: First submitted 2020-10-10; First posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) was considered as a heterogeneous disease with multi-organ and multi-system design, which is related to various complications, such as hypertension, obesity and arteriosclerosis. Ambulatory arterial stiffness index (AASI) is associated with arteriosclerosis and hypertension. There is no report on whether AASI is associated with left ventricular diastolic dysfunction in patients with HFpEF.

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction (HFpEF) is related to various complications, such as hypertension, obesity and arteriosclerosis. Ambulatory arterial stiffness index (AASI) is associated with arteriosclerosis and hypertension. AASI is especially associated with left ventricular diastolic dysfunction in patients with hypertension. Patients with HFpEF have obvious left ventricular diastolic insufficiency. However, there is still no research investigating the the relationship between AASI and left ventricular diastolic dysfunction in patients with HFpEF.

ELIGIBILITY:
Inclusion Criteria:

Adult aged >=18years old; Diagnosed with HFpEF.

Exclusion Criteria:

LVEF less than 45% at any time; Severe liver failure; Other causes of shortness of breath, such as severe pulmonary disease or severe Severe valvular disease of the left heart; Chronically bedridden or incapacitated; Age <18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients with preserved ejection fraction (HFpEF)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Left ventricular diastolic function | 1 day On admission
  the ratio of mitral peak velocity of early filling to early diastolic mitral annular velocity(E/e')

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No